CLINICAL TRIAL: NCT06446063
Title: Efficacy and Tolerance of the Cosmetic Care Product RV5098A on the Maintenance of Pigmentation on Face in Adult Patients With Vitiligo.
Brief Title: Efficacy & Tolerance of Cosmetic Product RV5098A on Face Pigmentation Maintenance in Adult Vitiligo Patients.
Status: Recruiting | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV5098A20230158
Record Dates: First submitted 2024-05-07; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Vitiligo
Keywords: Vitiligo; Adults; Face; Repigmented; Maintenance of repigmentation
MeSH Terms: conditions — Vitiligo; Facies | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated group
  Interventions: Other: Test product
- Control group
  Interventions: Other: Control Product

INTERVENTIONS:
Other: Test product — Twice daily applications The product is applied to the entire face.
  Groups: Treated group
Other: Control Product — Twice daily applications The product is applied to the entire face.
  Groups: Control group

SUMMARY:
Vitiligo is an autoimmune depigmentation disorder affecting 0.5 to 1% of the population worldwide. Vitiligo lesions are characterized by a progressive loss of pigmentation caused by the disappearance of functioning melanocytes in the epidermis, mainly resulting from the activation of immune cells in a genetically predisposed patient.

Despite major advances in the understanding of the mechanisms of the disease, the treatment remains challenging. Different treatment strategies could lead to cosmetically acceptable repigmentation (>75%), particularly on face and neck. However, after repigmentation, the risk of relapse is estimated at nearly 40% during the first year after stopping treatment.

To date, long-term management remains a challenge. With their topical product RV5098A adapted for patients with vitiligo, Pierre Fabre Laboratories hypothesize that it could be effective in maintaining pigmentation of previously repigmented lesions in adults with facial vitiligo.

ELIGIBILITY:
Inclusion Criteria:

Criteria related to the population:

- Subject aged between 18 and 75 years included.

Criteria related to the disease:

* Subject with facial vitiligo, regardless of its duration.
* having a sufficient repigmentation rate of the vitiligo after repigmenting treatment

Criteria related to treatments and/or products:

- Subject responder to a repigmenting treatment

Non-inclusion Criteria:

Criteria related to the diseases / skin condition:

* Subject with active vitiligo.
* Subject with spontaneous repigmentation without treatment.
* Subject having other dermatological condition, an acute, chronic, or progressive disease or history of disease liable to interfere with the study assessments or considered by the Investigator hazardous for the subject or incompatible with the study requirements.

Criteria related to treatments and/or products:

* Systemic immunomodulatory treatment taken for another pathology, before inclusion, on-going or planned to be established during the study.
* Any topical immunomodulatory treatment applied on the face for another pathology, on-going or planned to be established during the study.
* Any other topical or systemic treatment established or modified during the previous weeks or planned to be established or modified during the study, liable to interfere with the evaluation of the efficacy according to the investigator's assessment.
* Any dietary supplement for vitiligo within 4 weeks before the inclusion visit or planned to be established during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled from the investigator's outpatient's reception and/or from the database of the centre. The subjects corresponding to eligibility criteria may receive a phone call, a letter or an e-mail proposing to participate to the clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the test product RV5098A on the maintenance of pigmentation by the global evolution of facial vitiligo | assessed after 24 weeks of use
  assessed by the investigator on the face on a 7-point scale (from significant worsening to significant improvement)

SECONDARY OUTCOMES:
Efficacy of the test product RV5098A on the maintenance of pigmentation by the global evolution of facial vitiligo assessed by the investigator | assessed after 12 weeks of use
  assessed by the investigator on the face on a 7-point scale (from significant worsening to significant improvement)
Efficacy of the test product RV5098A on the maintenance of pigmentation by the global evolution of facial vitiligo assessed by the subject | assessed after 12 and 24 weeks of use and monthly at home
  assessed by the subject on the face on a 7-point scale (from very much worse to very much improved)
Efficacy of the test product RV5098A on the maintenance of pigmentation by the severity of facial vitiligo by the investigator | assessed at baseline and after 12 and 24 weeks of use.
  assessed by the investigator on the face on a vitiligo severity scale from 0 (absent) to 3 (complete depigmentation)
Efficacy of the test product RV5098A on the maintenance of pigmentation by the extent of facial vitiligo | assessed at baseline and after 12 and 24 weeks of use.
  assessed by the investigator on the face with score of extent of vitiligo
Efficacy of the test product RV5098A on the maintenance of pigmentation by the severity of facial vitiligo by the subject | assessed at baseline, after 12 and 24 weeks of use and monthly at home
  assessed by the subject on the face on a 5-point scale (from no vitiligo to very severe)
Efficacy of the test product RV5098A on the maintenance of pigmentation by the impact on quality of life assessed by the patient | assessed at baseline, after 12 and 24 weeks of use
  assessed by the subject with quality-of-life questionnaire
Efficacy of the test product RV5098A on the maintenance of pigmentation by imaging quantification. | assessed at baseline, after 12 and 24 weeks of use.
  Measurement of depigmentation surface on a target lesion of the face by the investigator.
Cosmetic satisfaction and perceived effects as regards to the use of the test product RV5098A by Cosmetic acceptability questionnaire assessed by the patient | assessed after 12 and 24 weeks of use.
  A questionnaire with a scale from 0 to 10 responding to statements about the sensorial experience and effect of the product (0=not at all agree, 10=completely agree).
Global tolerance of the test product RV5098A assessed by the investigator. | assessed after 24 weeks of use.
  assessed by the investigator with 5-point scale (from bad to excellent)
Compliance of the subjects to the test product RV5098A | through study completion, 6 months
  The subject will report his/her compliance in a subject's diary

CONTACTS AND LOCATIONS:
Overall Officials: Julien SENESCHAL, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- COSDERMA, Bordeaux, Gironde, France

IPD SHARING:
Plan to Share IPD: No